CLINICAL TRIAL: NCT01844505
Title: A Phase 3, Randomized, Double-Blind Study of Nivolumab Monotherapy or Nivolumab Combined With Ipilimumab Versus Ipilimumab Monotherapy in Subjects With Previously Untreated Unresectable or Metastatic Melanoma
Brief Title: Phase 3 Study of Nivolumab or Nivolumab Plus Ipilimumab Versus Ipilimumab Alone in Previously Untreated Advanced Melanoma (CheckMate 067)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA209-067; 2012-005371-13 (EudraCT Number)
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Unresectable or Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Nivolumab+Placebo for Ipilimumab+Placebo for Nivolumab (Experimental): Nivolumab 3 mg/kg solution intravenously every 2 weeks plus Placebo matching with Ipilimumab 0 mg/kg solution intravenously on weeks 1, 4 and Placebo matching with Nivolumab on weeks 4 for cycles 1 and 2, until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Interventions: Biological: Nivolumab; Biological: Placebo for Nivolumab; Biological: Placebo for Ipilimumab
- Arm B: Nivolumab+Ipilimumab+Placebo for Nivolumab (Experimental): Nivolumab 1 mg/kg solution intravenously combined with Ipilimumab 3 mg/kg solution intravenously every 3 weeks for 4 doses then Nivolumab 3 mg/kg solution intravenously every 2 weeks plus Placebo matching with Nivolumab on weeks 3 and 5 for cycles 1 and 2, until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Interventions: Biological: Nivolumab; Biological: Ipilimumab; Biological: Placebo for Nivolumab
- Arm C: Ipilimumab+Placebo for Nivolumab (Experimental): Ipilimumab 3 mg/kg solution intravenously every 3 weeks for a total of 4 doses plus Placebo matching with Nivolumab 0 mg/kg solution intravenously on weeks 3 and 5 for cycles 1 and 2, until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends (Placebo matching with Nivolumab is no longer required)
  Interventions: Biological: Ipilimumab; Biological: Placebo for Nivolumab

INTERVENTIONS:
Biological: Nivolumab
  Other Names: BMS-936558; MDX-1106
  Arms: Arm A: Nivolumab+Placebo for Ipilimumab+Placebo for Nivolumab; Arm B: Nivolumab+Ipilimumab+Placebo for Nivolumab
Biological: Ipilimumab
  Other Names: Yervoy; BMS-734016; MDX-010
  Arms: Arm B: Nivolumab+Ipilimumab+Placebo for Nivolumab; Arm C: Ipilimumab+Placebo for Nivolumab
Biological: Placebo for Nivolumab
Biological: Placebo for Ipilimumab
  Arms: Arm A: Nivolumab+Placebo for Ipilimumab+Placebo for Nivolumab

SUMMARY:
The purpose of this study is to show that Nivolumab and/or Nivolumab in combination with Ipilimumab will extend progression free survival and overall survival compared to Ipilimumab alone.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histologically confirmed stage III (unresectable) or stage IV melanoma
* Treatment naïve patients
* Measurable disease by computed tomography (CT) or Magnetic Resonance Imaging (MRI) per RECIST 1.1 criteria
* Tumor tissue from an unresectable or metastatic site of disease for biomarker analyses
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1

Exclusion Criteria:

* Active brain metastases or leptomeningeal metastases
* Ocular melanoma
* Subjects with active, known or suspected autoimmune disease
* Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of treatment
* Prior treatment with an anti-Programmed Death receptor-1 (PD-1), anti-Programmed Death-1 ligand-1 (PD-L1), anti-PD-L2, or anti-cytotoxic T lymphocyte associated antigen-4 (anti-CTLA-4) antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 945 (Actual)
Dates: Start 2013-06-11 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2024-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (150):
- United States (46):
  - Local Institution - 0085, Gilbert, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - Local Institution - 0046, La Jolla, California
  - Local Institution - 0053, Los Angeles, California
  - Local Institution - 0014, Los Angeles, California
  - Comprehensive Cancer Center At Desert Regional Medical Ctr, Palm Springs, California
  - Local Institution - 0066, Rancho Mirage, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - Local Institution - 0049, San Francisco, California
  - Local Institution - 0052, Aurora, Colorado
  - Local Institution - 0084, New Haven, Connecticut
  - Local Institution - 0098, Washington D.C., District of Columbia
  - Local Institution - 0183, Washington D.C., District of Columbia
  - Local Institution - 0042, Jacksonville, Florida
  - Local Institution - 0008, Orlando, Florida
  - Local Institution - 0051, Atlanta, Georgia
  - Maine Center For Cancer Medicine, Scarborough, Maine
  - Local Institution - 0080, Lutherville, Maryland
  - Local Institution - 0081, Boston, Massachusetts
  - Local Institution - 0082, Boston, Massachusetts
  - Local Institution - 0083, Boston, Massachusetts
  - Local Institution - 0087, Ann Arbor, Michigan
  - Local Institution - 0187, Minneapolis, Minnesota
  - Local Institution - 0065, Jackson, Mississippi
  - Local Institution - 0067, St Louis, Missouri
  - Local Institution - 0015, Las Vegas, Nevada
  - Local Institution - 0188, Morristown, New Jersey
  - Local Institution - 0068, Albuquerque, New Mexico
  - Local Institution - 0079, Albany, New York
  - Local Institution - 0174, New York, New York
  - Local Institution - 0070, New York, New York
  - Local Institution - 0047, Charlotte, North Carolina
  - Local Institution - 0048, Durham, North Carolina
  - Local Institution - 0007, Cleveland, Ohio
  - Local Institution - 0045, Portland, Oregon
  - Local Institution - 0061, Allentown, Pennsylvania
  - Local Institution - 0112, Bethlehem, Pennsylvania
  - Local Institution - 0069, Pittsburgh, Pennsylvania
  - Local Institution - 0154, Greenville, South Carolina
  - Local Institution - 0062, Nashville, Tennessee
  - Local Institution - 0064, Nashville, Tennessee
  - Local Institution - 0044, Dallas, Texas
  - Texas Oncology, Dallas, Texas
  - Local Institution - 0088, Houston, Texas
  - Local Institution - 0089, Salt Lake City, Utah
  - Local Institution - 0054, Seattle, Washington
- Australia (14):
  - Local Institution - 0017, Camperdown, New South Wales
  - Local Institution - 0031, Coffs Harbour, New South Wales
  - Local Institution - 0028, Gateshead, New South Wales
  - Local Institution - 0023, Macquarie University, New South Wales
  - Local Institution - 0138, North Sydney, New South Wales
  - Local Institution - 0019, Brisbane, Queensland
  - Local Institution - 0022, Southport, Queensland
  - Local Institution - 0018, Woolloongabba, Queensland
  - Local Institution - 0020, Adelaide, South Australia
  - Local Institution - 0025, Kurralta Park, South Australia
  - Local Institution - 0024, Box Hill, Victoria
  - Local Institution - 0016, Heidelberg, Victoria
  - Local Institution - 0026, Melbourne, Victoria
  - Local Institution - 0021, Nedlands, Western Australia
- Austria (2):
  - Local Institution - 0148, Salzburg
  - Local Institution - 0145, Vienna
- Belgium (5):
  - Local Institution - 0003, Brussels
  - Local Institution - 0002, Brussels
  - Local Institution - 0004, Edegem
  - Local Institution - 0005, Ghent
  - Local Institution - 0103, Leuven
- Canada (7):
  - Local Institution - 0140, Edmonton, Alberta
  - Local Institution - 0165, Vancouver, British Columbia
  - Local Institution - 0141, London, Ontario
  - Local Institution - 0143, Ottawa, Ontario
  - Local Institution - 0166, Toronto, Ontario
  - Local Institution - 0139, Montreal, Quebec
  - Local Institution - 0142, Québec, Quebec
- Czechia (4):
  - Local Institution - 0092, Brno
  - Local Institution - 0091, Hradec Králové
  - Local Institution - 0090, Prague
  - Local Institution - 0167, Prague
- Denmark (3):
  - Local Institution - 0076, Aarhus
  - Local Institution - 0078, Herlev
  - Local Institution - 0077, Odense
- Finland (2):
  - Local Institution - 0071, Helsinki, Uusimaa
  - Local Institution - 0169, Tampere
- France (7):
  - Local Institution - 0125, Boulogne-Billancourt
  - Local Institution - 0126, Marseille
  - Local Institution - 0056, Nantes
  - Local Institution - 0058, Paris
  - Local Institution - 0124, Pierre-Bénite
  - Local Institution - 0127, Rennes
  - Local Institution, Villejuif
- Germany (10):
  - Local Institution - 0162, Buxtehude
  - Local Institution - 0161, Erfurt
  - Local Institution - 0171, Erlangen
  - Local Institution - 0156, Essen
  - Local Institution - 0159, Hanover
  - Local Institution - 0157, Heidelberg
  - Local Institution - 0158, Kiel
  - Local Institution - 0178, Leipzig
  - Local Institution - 0160, München
  - Local Institution - 0134, Tübingen
- Ireland (6):
  - Local Institution - 0035, Dublin, Dublin
  - Local Institution - 0033, Cork
  - Local Institution - 0168, Dublin
  - Local Institution - 0036, Dublin
  - Local Institution - 0034, Dublin
  - Local Institution - 0032, Galway
- Israel (2):
  - Local Institution - 0120, Jerusalem
  - Local Institution - 0121, Tel Litwinsky
- Italy (9):
  - Local Institution - 0176, Bergamo
  - Local Institution - 0115, Genova
  - Local Institution - 0113, Meldola (FC)
  - Local Institution - 0172, Milan
  - Local Institution - 0117, Milan
  - Local Institution - 0114, Napoli
  - Local Institution - 0118, Padua
  - Local Institution - 0177, Roma
  - Local Institution - 0116, Siena
- Netherlands (3):
  - Local Institution - 0010, Amsterdam
  - Local Institution - 0012, Leiden
  - Local Institution - 0013, Nijmegen
- Local Institution - 0029, Auckland, New Zealand
- Local Institution - 0123, Oslo, Norway
- Poland (4):
  - Local Institution - 0109, Gdansk
  - Local Institution - 0133, Krakow
  - Local Institution - 0060, Lodz
  - Local Institution - 0059, Warsaw
- Russia (4):
  - Local Institution - 0130, Moscow
  - Local Institution - 0132, Saint Petersburg
  - Local Institution - 0128, Saint Petersburg
  - Local Institution - 0131, Samara
- Spain (7):
  - Local Institution - 0152, Badalona-Barcelona
  - Local Institution - 0151, Barcelona
  - Local Institution - 0175, Barcelona
  - Local Institution - 0150, Madrid
  - Local Institution - 0149, Madrid
  - Local Institution - 0153, Málaga
  - Local Institution - 0147, Pamplona
- Sweden (2):
  - Local Institution - 0182, Gothenberg
  - Local Institution - 0184, Stockholm
- Switzerland (4):
  - Local Institution - 0164, Geneva
  - Local Institution - 0189, Lausanne
  - Local Institution - 0186, Sankt Gallen
  - Local Institution - 0163, Zurich
- United Kingdom (7):
  - Local Institution - 0039, Glasgow, Dumfries & Galloway
  - Local Institution - 0038, London, Greater London
  - Local Institution - 0119, Manchester, Greater Manchester
  - Local Institution - 0041, Northwood, Middlesex
  - Local Institution - 0122, Nottingham, Nottinghamshire
  - Local Institution - 0037, Cambridge
  - Local Institution - 0040, Swansea

REFERENCES:
- [Derived] Long GV, Larkin J, Schadendorf D, Grob JJ, Lao CD, Marquez-Rodas I, Wagstaff J, Lebbe C, Pigozzo J, Robert C, Ascierto PA, Atkinson V, Postow MA, Atkins MB, Sznol M, Callahan MK, Topalian SL, Sosman JA, Kotapati S, Thakkar PK, Ritchings C, Pe Benito M, Re S, Soleymani S, Hodi FS. Pooled Long-Term Outcomes With Nivolumab Plus Ipilimumab or Nivolumab Alone in Patients With Advanced Melanoma. J Clin Oncol. 2025 Mar 10;43(8):938-948. doi: 10.1200/JCO.24.00400. Epub 2024 Nov 6. PMID 39504507
- [Derived] Wolchok JD, Chiarion-Sileni V, Rutkowski P, Cowey CL, Schadendorf D, Wagstaff J, Queirolo P, Dummer R, Butler MO, Hill AG, Postow MA, Gaudy-Marqueste C, Medina T, Lao CD, Walker J, Marquez-Rodas I, Haanen JBAG, Guidoboni M, Maio M, Schoffski P, Carlino MS, Sandhu S, Lebbe C, Ascierto PA, Long GV, Ritchings C, Nassar A, Askelson M, Benito MP, Wang W, Hodi FS, Larkin J; CheckMate 067 Investigators. Final, 10-Year Outcomes with Nivolumab plus Ipilimumab in Advanced Melanoma. N Engl J Med. 2025 Jan 2;392(1):11-22. doi: 10.1056/NEJMoa2407417. Epub 2024 Sep 15. PMID 39282897
- [Derived] Mantia CM, Werner L, Stwalley B, Ritchings C, Tarhini AA, Atkins MB, McDermott DF, Regan MM. Sensitivity of treatment-free survival to subgroup analyses in patients with advanced melanoma treated with immune checkpoint inhibitors. Melanoma Res. 2022 Feb 1;32(1):35-44. doi: 10.1097/CMR.0000000000000793. PMID 34855329
- [Derived] Wolchok JD, Chiarion-Sileni V, Gonzalez R, Grob JJ, Rutkowski P, Lao CD, Cowey CL, Schadendorf D, Wagstaff J, Dummer R, Ferrucci PF, Smylie M, Butler MO, Hill A, Marquez-Rodas I, Haanen JBAG, Guidoboni M, Maio M, Schoffski P, Carlino MS, Lebbe C, McArthur G, Ascierto PA, Daniels GA, Long GV, Bas T, Ritchings C, Larkin J, Hodi FS. Long-Term Outcomes With Nivolumab Plus Ipilimumab or Nivolumab Alone Versus Ipilimumab in Patients With Advanced Melanoma. J Clin Oncol. 2022 Jan 10;40(2):127-137. doi: 10.1200/JCO.21.02229. Epub 2021 Nov 24. PMID 34818112
- [Derived] Larkin J, Chiarion-Sileni V, Gonzalez R, Grob JJ, Rutkowski P, Lao CD, Cowey CL, Schadendorf D, Wagstaff J, Dummer R, Ferrucci PF, Smylie M, Hogg D, Hill A, Marquez-Rodas I, Haanen J, Guidoboni M, Maio M, Schoffski P, Carlino MS, Lebbe C, McArthur G, Ascierto PA, Daniels GA, Long GV, Bastholt L, Rizzo JI, Balogh A, Moshyk A, Hodi FS, Wolchok JD. Five-Year Survival with Combined Nivolumab and Ipilimumab in Advanced Melanoma. N Engl J Med. 2019 Oct 17;381(16):1535-1546. doi: 10.1056/NEJMoa1910836. Epub 2019 Sep 28. PMID 31562797
- [Derived] Hodi FS, Chiarion-Sileni V, Gonzalez R, Grob JJ, Rutkowski P, Cowey CL, Lao CD, Schadendorf D, Wagstaff J, Dummer R, Ferrucci PF, Smylie M, Hill A, Hogg D, Marquez-Rodas I, Jiang J, Rizzo J, Larkin J, Wolchok JD. Nivolumab plus ipilimumab or nivolumab alone versus ipilimumab alone in advanced melanoma (CheckMate 067): 4-year outcomes of a multicentre, randomised, phase 3 trial. Lancet Oncol. 2018 Nov;19(11):1480-1492. doi: 10.1016/S1470-2045(18)30700-9. Epub 2018 Oct 22. PMID 30361170
- [Derived] Wolchok JD, Chiarion-Sileni V, Gonzalez R, Rutkowski P, Grob JJ, Cowey CL, Lao CD, Wagstaff J, Schadendorf D, Ferrucci PF, Smylie M, Dummer R, Hill A, Hogg D, Haanen J, Carlino MS, Bechter O, Maio M, Marquez-Rodas I, Guidoboni M, McArthur G, Lebbe C, Ascierto PA, Long GV, Cebon J, Sosman J, Postow MA, Callahan MK, Walker D, Rollin L, Bhore R, Hodi FS, Larkin J. Overall Survival with Combined Nivolumab and Ipilimumab in Advanced Melanoma. N Engl J Med. 2017 Oct 5;377(14):1345-1356. doi: 10.1056/NEJMoa1709684. Epub 2017 Sep 11. PMID 28889792
- [Derived] Long GV, Weber JS, Larkin J, Atkinson V, Grob JJ, Schadendorf D, Dummer R, Robert C, Marquez-Rodas I, McNeil C, Schmidt H, Briscoe K, Baurain JF, Hodi FS, Wolchok JD. Nivolumab for Patients With Advanced Melanoma Treated Beyond Progression: Analysis of 2 Phase 3 Clinical Trials. JAMA Oncol. 2017 Nov 1;3(11):1511-1519. doi: 10.1001/jamaoncol.2017.1588. PMID 28662232
- [Derived] Schadendorf D, Larkin J, Wolchok J, Hodi FS, Chiarion-Sileni V, Gonzalez R, Rutkowski P, Grob JJ, Cowey CL, Lao C, Wagstaff J, Callahan MK, Postow MA, Smylie M, Ferrucci PF, Dummer R, Hill A, Taylor F, Sabater J, Walker D, Kotapati S, Abernethy A, Long GV. Health-related quality of life results from the phase III CheckMate 067 study. Eur J Cancer. 2017 Sep;82:80-91. doi: 10.1016/j.ejca.2017.05.031. Epub 2017 Jun 23. PMID 28651159
- [Derived] Larkin J, Chiarion-Sileni V, Gonzalez R, Grob JJ, Cowey CL, Lao CD, Schadendorf D, Dummer R, Smylie M, Rutkowski P, Ferrucci PF, Hill A, Wagstaff J, Carlino MS, Haanen JB, Maio M, Marquez-Rodas I, McArthur GA, Ascierto PA, Long GV, Callahan MK, Postow MA, Grossmann K, Sznol M, Dreno B, Bastholt L, Yang A, Rollin LM, Horak C, Hodi FS, Wolchok JD. Combined Nivolumab and Ipilimumab or Monotherapy in Untreated Melanoma. N Engl J Med. 2015 Jul 2;373(1):23-34. doi: 10.1056/NEJMoa1504030. Epub 2015 May 31. PMID 26027431
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab: Nivolumab monotherapy 3 mg/kg intravenous (IV) once every 2 weeks (Q2W) until disease progression or unacceptable toxicity
- Nivolumab + Ipilimumab: Nivolumab 1 mg/kg IV combined with Ipilimumab 3 mg/kg IV once every 3 weeks (Q3W) for 4 doses followed by nivolumab 3 mg/kg IV Q2W until disease progression or unacceptable toxicity
- Ipilimumab: Ipilimumab monotherapy 3 mg/kg IV Q3W for a total of 4 doses
Period: Pre-Treatment Period
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab
Started | 316 | 314 | 315
Completed | 313 | 313 | 311
Not Completed | 3 | 1 | 4
Period: Treatment Period
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab
Started | 313 | 313 | 311
Completed | 0 | 0 | 0
Not Completed | 313 | 313 | 311
Not completed — SUBJECT WITHDREW CONSENT | 9 | 12 | 19
Not completed — Other Reasons | 120 | 136 | 58
Not completed — Lost to Follow-up | 9 | 11 | 6
Not completed — Death | 175 | 154 | 228

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab | Total
Number analyzed (Participants) | 316 | 314 | 315 | 945
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (13.92) | 59.3 (13.86) | 60.8 (13.23) | 59.6 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 108 | 113 | 335
  Male | 202 | 206 | 202 | 610
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE | 308 | 310 | 303 | 921
  BLACK OR AFRICAN AMERICAN | 0 | 0 | 0 | 0
  ASIAN | 2 | 2 | 6 | 10
  AMERICAN INDIAN OR ALASKA NATIVE | 1 | 0 | 0 | 1
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 1 | 0 | 0 | 1
  OTHER | 4 | 2 | 5 | 11
  NOT REPORTED | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time between the date of randomization and the first date of documented progression, as determined by the Investigator, or death due to any cause, whichever occurred first. Participants who died without a reported progression were considered to have progressed on the date of their death. Participants who did not progress or die were censored on the date of their last evaluable tumor assessment. Participants who did not have any on study tumor assessments and did not die were censored on their date of randomization. Participants treated beyond progression were considered to have progressive disease at the time of the initial progression event regardless of subsequent tumor response. Particpants who started anti-cancer therapy without a prior reported progression were censored on the date of their last evaluable tumor assessment prior to the initiation of subsequent anti-cancer therapy.
Time Frame: From randomization until disease progression or death, whichever occurred first (assessed up to February 2015, approximately 20 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 316 | 314 | 315
months | 6.87 [4.34 to 9.46] | 11.50 [8.90 to 16.72] | 2.89 [2.79 to 3.42]
Statistical Analysis 1: Comparison: Nivolumab vs Ipilimumab; Test type: Superiority or Other; p < 0.0001, Stratified Log Rank test; Hazard Ratio (HR) = 0.57, 99.5% CI 2-sided [0.43 to 0.76] — Stratified Cox proportional hazard model. Ratio of Nivolumab over Ipimlimumab
Statistical Analysis 2: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority or Other; p < 0.0001, Stratified Log Rank test; Hazard Ratio (HR) = 0.42, 99.5% CI 2-sided [0.31 to 0.57] — Stratified Cox proportional hazard model. Ratio of Nivolumab+Ipilimumab over Ipilimumab

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time between the date of randomization and the date of death. For participants without documentation of death, OS was censored on the last date the participant was known to be alive.
Time Frame: From randomization to date of death (Assessed up to September 2016, approximately 39 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 316 | 314 | 315
months | NA [29.08 to NA] — Median OS was not reached | NA [NA to NA] — Median OS was not reached | 19.98 [17.08 to 24.61]
Statistical Analysis 1: Comparison: Nivolumab vs Ipilimumab; Test type: Superiority or Other; p < 0.0001, Log Rank; Log-rank Test stratified by PD-L1 status, BRAF status, and M stage at screening as entered into the Interactive Voice Response System (IVRS); Hazard Ratio (HR) = 0.63, 98% CI 2-sided [0.50 to 0.78] — Stratified Cox proportional hazard model. Ratio of Nivolumab over Ipilimumab
Statistical Analysis 2: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority or Other; p < 0.0001, Log Rank; Log-rank Test stratified by PD-L1 status, BRAF status, and M stage at screening as entered into the IVRS; Hazard Ratio (HR) = 0.55, 98% CI 2-sided [0.42 to 0.72] — Stratified Cox proportional hazard model. Ratio of Nivolumab+Ipilimumab over Ipilimumab

3. Primary Outcome: Rate of Overall Survival
Description: OS was defined as the time between the date of randomization and the date of death. For participants without documentation of death, OS was censored on the last date the participant was known to be alive. The overall survival rate at time T (6, 12, or 24 months) was defined as the probability that a participant was alive at time T following randomization.
Time Frame: 24 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Probability of survival at Time T
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 316 | 314 | 315
Probability of survival at Time T
  Rate of OS at 6 months | 0.85 [0.81 to 0.89] | 0.86 [0.81 to 0.89] | 0.82 [0.78 to 0.86]
  Rate of OS at 12 months | 0.74 [0.69 to 0.79] | 0.73 [0.68 to 0.78] | 0.67 [0.61 to 0.72]
  Rate of OS at 24 months | 0.59 [0.53 to 0.64] | 0.64 [0.59 to 0.69] | 0.45 [0.39 to 0.50]

4. Primary Outcome: Rate of Progression-Free Survival
Description: PFS was defined as the time between the date of randomization and the first date of documented progression, as determined by the Investigator, or death due to any cause, whichever occurred first. Participants who died without a reported progression were considered to have progressed on the date of their death. Participants who did not progress or die were censored on the date of their last evaluable tumor assessment. Participants who did not have any on study tumor assessments and did not die were censored on their date of randomization. Participants treated beyond progression were considered to have progressive disease at the time of the initial progression event regardless of subsequent tumor response. Participants who started anti-cancer therapy without a prior reported progression were censored on the date of their last evaluable tumor assessment prior to the initiation of subsequent anti-cancer therapy.
Time Frame: 24 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 316 | 314 | 315
Percentage of participants
  Rate at 6 months | 0.52 [0.46 to 0.58] | 0.63 [0.57 to 0.68] | 0.28 [0.23 to 0.33]
  Rate at 12 months | 0.43 [0.37 to 0.49] | 0.50 [0.44 to 0.55] | 0.18 [0.14 to 0.22]
  Rate at 24 months | 0.37 [0.31 to 0.43] | 0.43 [0.37 to 0.48] | 0.12 [0.09 to 0.17]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: as for outcome 4
Time Frame: From randomization until disease progression or death, whichever occurred first (assessed up to approximately 128 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 316 | 314 | 315
months | 6.93 [5.13 to 10.18] | 11.50 [8.90 to 20.04] | 2.86 [2.79 to 3.09]
Statistical Analysis 1: Comparison: Nivolumab vs Nivolumab + Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.65 to 0.96] — Stratified Cox proportional hazard model. Hazard Ratio is Nivolumab + Ipilimumab over Nivolumab

6. Secondary Outcome: Overall Survival (OS)
Description: as for outcome 2
Time Frame: From randomization until death (assessed up to approximately 128 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 316 | 314 | 315
months | 36.93 [28.25 to 58.71] | 71.92 [38.18 to 114.37] | 19.94 [16.85 to 24.61]
Statistical Analysis 1: Comparison: Nivolumab vs Nivolumab + Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.69 to 1.05] — Stratified Cox proportional hazard model. Hazard Ratio is Nivolumab + Ipilimumab over Nivolumab

7. Secondary Outcome: Objective Response Rate (ORR) Per Investigator Assessment
Description: The ORR was defined as the percentage of participants with a best overall response (BOR) of a complete response (CR) or partial response (PR) divided by the number of randomized participants for each arm. The BOR was defined as the best response designation, as determined by the Investigator, recorded between the date of randomization and the date of progression, as assessed by the Investigator per RECIST 1.1 or the date of subsequent anticancer therapy (including tumor-directed radiotherapy and tumor-directed surgery), whichever occurred first. For participants without evidence of RECIST 1.1 progression or subsequent anticancer therapy, all available response designations contributed to the BOR assessment. CR= Disappearance of all evidence of disease, confirmed by PET scan; PR= Regression of measureable disease and no new sites; Stable Disease (SD)= Failure to attain CR/PR or PD; Progressive Disease (PD)= Any new lesion or increase by >=50% of previously involved sites from nadir.
Time Frame: as for outcome 5
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 316 | 314 | 315
Percentage of participants | 44.9 [39.4 to 50.6] | 58.3 [52.6 to 63.8] | 19.0 [14.9 to 23.8]
Statistical Analysis 1: Comparison: Nivolumab vs Ipilimumab; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.59, 95% CI 2-sided [2.49 to 5.16] — Cochran-Mantel-Haenszel Test Stratified by PD-L1 Status, BRAF Status and M stage at screening as entered into the IVRS. Ratio of Nivolumab over Ipilimumab
Statistical Analysis 2: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 6.35, 95% CI 2-sided [4.38 to 9.22] — Cochran-Mantel-Haenszel Test Stratified by PD-L1 Status, BRAF Status and M stage at screening as entered into the IVRS. Ratio of Nivolumab + Ipilimumab over Ipilimumab
Statistical Analysis 3: Comparison: Nivolumab vs Ipilimumab; Test type: Superiority or Other; Difference of Objective Response Rates = 26.0, 95% CI 2-sided [19.1 to 32.8] — Difference in ORR and corresponding 95% CI is based on Cochran-Mantel-Haenszel (CMH) method of weighting, adjusting for PD-L1 Status, BRAF Mutation Status and M-stage at screening as entered into the IVRS. Difference of Nivolumab - Ipilimumab
Statistical Analysis 4: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority or Other; Difference of Objective Response Rates = 39.0, 95% CI 2-sided [32.2 to 45.9] — Difference in ORR and corresponding 95% CI is based on CMH method of weighting, adjusting for PD-L1 Status, BRAF Mutation Status and M-stage at screening as entered into the IVRS. Difference of Nivolumab and Ipilimumab - Ipilimumab
Statistical Analysis 5: Comparison: Nivolumab vs Nivolumab + Ipilimumab; Test type: Superiority or Other; Odds Ratio (OR) = 1.75, 95% CI 2-sided [1.26 to 2.42] — Cochran-Mantel-Haenszel Test Stratified by PD-L1 Status, BRAF Status and M stage at screening as entered into the IVRS. Ratio of Nivolumab + Ipilimumab over Nivolumab
Statistical Analysis 6: Comparison: Nivolumab vs Nivolumab + Ipilimumab; Test type: Superiority or Other; Difference of Objective Response Rates = 13.2, 95% CI 2-sided [5.7 to 20.7] — Difference in ORR and corresponding 95% CI is based on CMH method of weighting, adjusting for PD-L1 Status, BRAF Mutation Status and M-stage at screening as entered into the IVRS. Difference of Nivolumab and Ipilimumab - Nivolumab

8. Secondary Outcome: Progression-Free Survival Based on PD-L1 Expression Level
Description: PD-L1 expression was defined as the percent of tumor cells demonstrating plasma membrane PD-L1 staining of any intensity using an IHC assay. Tumor biopsy specimens without measurable PD-L1 expression were classified as indeterminate if the staining was hampered for reasons attributed to the biology of the specimen and not because of improper specimen preparation or handling. Missing specimens, specimens that were not optimally collected (ie not evaluable), and all other specimens were classified as unknown. Participants must have been classified as PD-L1 >=5% or PD-L1 <5% per a verified IHC assay, or as indeterminate (ie not unknown), in order to be randomized.
Time Frame: From randomization until disease progression or death from any cause, whichever occurs first (Assessed up to September 2016, approximately 39 months)
Population: All randomized participants with evaluable PD-L1 expression level at baseline
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 316 | 314 | 315
months
  PD-L1 < 1% (n=117, 123, 113): number analyzed (Participants) | 117 | 123 | 113
  PD-L1 < 1% (n=117, 123, 113) | 2.83 [2.76 to 5.39] | 11.17 [6.93 to 26.68] | 2.76 [2.66 to 2.86]
  PD-L1 >= 1% (n= 171, 155, 164): number analyzed (Participants) | 171 | 155 | 164
  PD-L1 >= 1% (n= 171, 155, 164) | 16.20 [8.11 to 27.66] | 16.72 [9.72 to NA] — Upper 95% Confidence Interval was not reached. | 3.48 [2.83 to 4.17]
  PD-L1 < 5% (n= 208, 210, 202): number analyzed (Participants) | 208 | 210 | 202
  PD-L1 < 5% (n= 208, 210, 202) | 5.32 [2.96 to 6.87] | 11.17 [8.31 to 22.18] | 2.83 [2.76 to 3.02]
  PD-L1 >= 5% (n= 80, 68, 75): number analyzed (Participants) | 80 | 68 | 75
  PD-L1 >= 5% (n= 80, 68, 75) | 22.34 [9.46 to NA] — Upper 95% Confidence Interval was not reached. | 22.11 [9.72 to NA] — Upper 95% Confidence Interval was not reached. | 3.94 [2.79 to 4.21]
  PD-L1 < 10% (n= 229, 232, 223): number analyzed (Participants) | 229 | 232 | 223
  PD-L1 < 10% (n= 229, 232, 223) | 5.62 [3.09 to 8.87] | 11.10 [8.02 to 18.14] | 2.83 [2.76 to 3.02]
  PD-L1 >= 10% (n= 59, 46, 54): number analyzed (Participants) | 59 | 46 | 54
  PD-L1 >= 10% (n= 59, 46, 54) | 21.98 [9.07 to NA] — Upper 95% Confidence Interval was not reached. | NA [13.96 to NA] — Median and upper 95% Confidence Interval were not reached. | 4.11 [2.79 to 5.59]
  PD-L1 Indeterminate/ Not Evaluable (n= 28, 36, 38): number analyzed (Participants) | 28 | 36 | 38
  PD-L1 Indeterminate/ Not Evaluable (n= 28, 36, 38) | 2.99 [2.66 to 6.93] | 6.93 [2.79 to 20.04] | 2.83 [2.60 to 6.41]
Statistical Analysis 1: Comparison: Nivolumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.46 to 0.85] — HR of Nivolumab vs. Ipilimumab in participants with PD-L1 expression < 1%
Statistical Analysis 2: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.39, 95% CI 2-sided [0.28 to 0.54] — HR of Nivolumab+Ipilimumab vs. Ipilimumab in participants with PD-L1 expression < 1%
Statistical Analysis 3: Comparison: Nivolumab vs Nivolumab + Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.45 to 0.87] — HR of Nivolumab+Ipilimumab vs. Nivolumab in participants with PD-L1 expression < 1%
Statistical Analysis 4: Comparison: Nivolumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.34 to 0.59] — HR of Nivolumab vs. Ipilimumab in participants with PD-L1 expression >= 1%
Statistical Analysis 5: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.40, 95% CI 2-sided [0.30 to 0.53] — HR of Nivolumab+Ipilimumab vs. Ipilimumab in participants with PD-L1 expression >= 1%
Statistical Analysis 6: Comparison: Nivolumab vs Nivolumab + Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.66 to 1.21] — HR of Nivolumab+Ipilimumab vs. Nivolumab in participants with PD-L1 expression >= 1%
Statistical Analysis 7: Comparison: Nivolumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.45 to 0.71] — HR of Nivolumab vs. Ipilimumab in participants with PD-L1 expression < 5%
Statistical Analysis 8: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.33 to 0.53] — HR of Nivolumab+Ipilimumab vs. Ipilimumab in participants with PD-L1 expression < 5%
Statistical Analysis 9: Comparison: Nivolumab vs Nivolumab + Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.57 to 0.94] — HR of Nivolumab+Ipilimumab vs. Nivolumab in participants with PD-L1 expression < 5%
Statistical Analysis 10: Comparison: Nivolumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.40, 95% CI 2-sided [0.27 to 0.60] — HR of Nivolumab vs. Ipilimumab in participants with PD-L1 expression >= 5%
Statistical Analysis 11: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.22 to 0.54] — HR of Nivolumab+Ipilimumab vs. Ipilimumab in participants with PD-L1 expression >= 5%
Statistical Analysis 12: Comparison: Nivolumab vs Nivolumab + Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.54 to 1.38] — HR of Nivolumab+Ipilimumab vs. Nivolumab in participants with PD-L1 expression >= 5%
Statistical Analysis 13: Comparison: Nivolumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.43 to 0.67] — HR of Nivolumab vs. Ipilimumab in participants with PD-L1 expression < 10%
Statistical Analysis 14: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.34 to 0.54] — HR of Nivolumab+Ipilimumab vs. Ipilimumab in participants with PD-L1 expression < 10%
Statistical Analysis 15: Comparison: Nivolumab vs Nivolumab + Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.63 to 1.01] — HR of Nivolumab+Ipilimumab vs. Nivolumab in participants with PD-L1 expression < 10%
Statistical Analysis 16: Comparison: Nivolumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.28 to 0.73] — HR of Nivolumab vs. Ipilimumab in participants with PD-L1 expression >= 10%
Statistical Analysis 17: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.28, 95% CI 2-sided [0.16 to 0.49] — HR of Nivolumab+Ipilimumab vs. Ipilimumab in participants with PD-L1 expression >= 10%
Statistical Analysis 18: Comparison: Nivolumab vs Nivolumab + Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.34 to 1.09] — HR of Nivolumab+Ipilimumab vs. Nivolumab in participants with PD-L1 expression >= 10%
Statistical Analysis 19: Comparison: Nivolumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.49 to 1.52] — HR of Nivolumab vs. Ipilimumab in participants with PD-L1 expression not evaluable at baseline
Statistical Analysis 20: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.30 to 0.89] — HR of Nivolumab+Ipilimumab vs. Ipilimumab in participants with PD-L1 expression not evaluable at baseline
Statistical Analysis 21: Comparison: Nivolumab vs Nivolumab + Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.33 to 1.09] — HR of Nivolumab+Ipilimumab vs. Nivolumab in participants with PD-L1 expression not evaluable at baseline

9. Secondary Outcome: Overall Survival Based on PD-L1 Expression Level
Description: as for outcome 2
Time Frame: From randomization until death (assessed up to approximately 128 months)
Population: All randomized participants with evaluable PD-L1 expression level at baseline
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 316 | 314 | 315
months
  PD-L1 < 1% (n=117, 123, 113): number analyzed (Participants) | 117 | 123 | 113
  PD-L1 < 1% (n=117, 123, 113) | 23.46 [13.01 to NA] — Upper 95% Confidence Interval was not reached | NA [26.45 to NA] — Upper 95% Confidence Interval was not reached | 18.56 [13.67 to 23.20]
  PD-L1 >= 1% (n= 171, 155, 164): number analyzed (Participants) | 171 | 155 | 164
  PD-L1 >= 1% (n= 171, 155, 164) | 85.09 [39.00 to NA] — Upper 95% Confidence Interval was not reached | 82.30 [39.06 to NA] — Upper 95% Confidence Interval was not reached | 21.49 [16.85 to 29.08]
  PD-L1 < 5% (n= 208, 210, 202): number analyzed (Participants) | 208 | 210 | 202
  PD-L1 < 5% (n= 208, 210, 202) | 35.94 [23.06 to 59.24] | 65.94 [32.72 to 114.37] | 18.40 [13.70 to 22.51]
  PD-L1 >= 5% (n= 80, 68, 75): number analyzed (Participants) | 80 | 68 | 75
  PD-L1 >= 5% (n= 80, 68, 75) | 64.51 [33.64 to NA] — Upper 95% Confidence Interval was not reached | 104.97 [39.06 to NA] — Upper 95% Confidence Interval was not reached | 28.88 [18.10 to 44.16]
  PD-L1 < 10% (n= 229, 232, 223): number analyzed (Participants) | 229 | 232 | 223
  PD-L1 < 10% (n= 229, 232, 223) | 36.93 [23.46 to 80.85] | 70.74 [34.83 to 107.89] | 18.56 [14.98 to 23.03]
  PD-L1 >= 10% (n= 59, 46, 54): number analyzed (Participants) | 59 | 46 | 54
  PD-L1 >= 10% (n= 59, 46, 54) | 43.63 [31.24 to NA] — Upper 95% Confidence Interval was not reached | NA [39.06 to NA] — Upper 95% Confidence Interval was not reached | 29.08 [17.45 to 46.55]
  PD-L1 Indeterminate/ Not Evaluable (n= 28, 36, 38): number analyzed (Participants) | 28 | 36 | 38
  PD-L1 Indeterminate/ Not Evaluable (n= 28, 36, 38) | 23.89 [11.76 to NA] — Upper 95% Confidence Interval was not reached | NA [21.39 to NA] — Median and Upper 95% Confidence Interval were not reached | 18.73 [8.41 to 30.00]
Statistical Analysis 1: Comparison: Nivolumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.57 to 1.05] — HR of Nivolumab vs. Ipilimumab in participants with PD-L1 expression < 1%
Statistical Analysis 2: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.43 to 0.81] — HR of Nivolumab+Ipilimumab vs. Ipilimumab in participants with PD-L1 expression < 1%
Statistical Analysis 3: Comparison: Nivolumab vs Nivolumab + Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.76, 95% CI [0.55 to 1.04] — HR of Nivolumab+Ipilimumab vs. Nivolumab in participants with PD-L1 expression < 1%
Statistical Analysis 4: Comparison: Nivolumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.39 to 0.68] — HR of Nivolumab vs. Ipilimumab in participants with PD-L1 expression >= 1%
Statistical Analysis 5: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.38 to 0.67] — HR of Nivolumab+Ipilimumab vs. Ipilimumab in participants with PD-L1 expression >= 1%
Statistical Analysis 6: Comparison: Nivolumab vs Nivolumab + Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.72 to 1.31] — HR of Nivolumab+Ipilimumab vs. Nivolumab in participants with PD-L1 expression >= 1%
Statistical Analysis 7: Comparison: Nivolumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.49 to 0.78] — HR of Nivolumab vs. Ipilimumab in participants with PD-L1 expression < 5%
Statistical Analysis 8: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.41 to 0.66] — HR of Nivolumab+Ipilimumab vs. Ipilimumab in participants with PD-L1 expression < 5%
Statistical Analysis 9: Comparison: Nivolumab vs Nivolumab + Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.66 to 1.08] — HR of Nivolumab+Ipilimumab vs. Nivolumab in participants with PD-L1 expression < 5%
Statistical Analysis 10: Comparison: Nivolumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.41 to 0.91] — HR of Nivolumab vs. Ipilimumab in participants with PD-L1 expression >= 5%
Statistical Analysis 11: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.38 to 0.91] — HR of Nivolumab+Ipilimumab vs. Ipilimumab in participants with PD-L1 expression >= 5%
Statistical Analysis 12: Comparison: Nivolumab vs Nivolumab + Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.62 to 1.53] — HR of Nivolumab+Ipilimumab vs. Nivolumab in participants with PD-L1 expression >= 5%
Statistical Analysis 13: Comparison: Nivolumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.48 to 0.75] — HR of Nivolumab vs. Ipilimumab in participants with PD-L1 expression < 10%
Statistical Analysis 14: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.43 to 0.68] — HR of Nivolumab+Ipilimumab vs. Ipilimumab in participants with PD-L1 expression < 10%
Statistical Analysis 15: Comparison: Nivolumab vs Nivolumab + Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.71 to 1.14] — HR of Nivolumab+Ipilimumab vs. Nivolumab in participants with PD-L1 expression < 10%
Statistical Analysis 16: Comparison: Nivolumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.44 to 1.10] — HR of Nivolumab vs. Ipilimumab in participants with PD-L1 expression >= 10%
Statistical Analysis 17: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.32 to 0.91] — HR of Nivolumab+Ipilimumab vs. Ipilimumab in participants with PD-L1 expression >= 10%
Statistical Analysis 18: Comparison: Nivolumab vs Nivolumab + Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.45 to 1.32] — HR of Nivolumab+Ipilimumab vs. Nivolumab in participants with PD-L1 expression >= 10%
Statistical Analysis 19: Comparison: Nivolumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.37 to 1.34] — HR of Nivolumab vs. Ipilimumab in participants with PD-L1 expression not evaluable at baseline
Statistical Analysis 20: Comparison: Nivolumab + Ipilimumab vs Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.26 to 0.91] — HR of Nivolumab+Ipilimumab vs. Ipilimumab in participants with PD-L1 expression not evaluable at baseline
Statistical Analysis 21: Comparison: Nivolumab vs Nivolumab + Ipilimumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.34 to 1.39] — HR of Nivolumab+Ipilimumab vs. Nivolumab in participants with PD-L1 expression not evaluable at baseline

10. Secondary Outcome: Mean Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Global Health Status
Description: Health Related Quality of Life was assessed using the EORTC QLQ-C30 questionnaire Version 3. With the exception of 2 items included in the global health/quality of life scale, for which responses range from 1 (Very poor) to 7 (Excellent), item responses range from 1 (Not at all) to 4 (Very much). Raw scores for the EORTC QLQ-C30 are transformed to a 0-100 metric such that higher scores for all functional scales and Global Health Status indicate better HRQoL; an increase from baseline indicates improvement in HRQoL compared to baseline.
Time Frame: Baseline (Day 1) and Week 5, 7, 11, 13, 17, 19, 23, 25, 31, 37, 43, 49, 55, 61, 67, 73, 79, 85, 91, 97, 103, 109, 115, 121, 127, 133, 139, 145, 151 and 157
Population: All randomized participants. Only participants with evaluable EORTC scores at baseline and at particular timepoint are considered in the analysis.
Measure: Mean (Standard Deviation); unit: Points on EORTC scale
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 316 | 314 | 315
Points on EORTC scale
  Week 5 (n= 233, 183, 221): number analyzed (Participants) | 233 | 183 | 221
  Week 5 (n= 233, 183, 221) | -2.8 (15.74) | -4.3 (21.38) | -3.1 (17.24)
  Week 7 (n= 239, 183, 218): number analyzed (Participants) | 239 | 183 | 218
  Week 7 (n= 239, 183, 218) | -2.6 (16.89) | -5.0 (20.60) | -4.3 (18.07)
  Week 11 (n= 201, 112, 163): number analyzed (Participants) | 201 | 112 | 163
  Week 11 (n= 201, 112, 163) | -2.0 (18.10) | -2.4 (21.99) | -6.2 (18.73)
  Week 13 (n= 195, 106, 130): number analyzed (Participants) | 195 | 106 | 130
  Week 13 (n= 195, 106, 130) | -1.9 (16.44) | -3.8 (21.21) | -5.5 (20.27)
  Week 17 (n= 158, 84, 104): number analyzed (Participants) | 158 | 84 | 104
  Week 17 (n= 158, 84, 104) | -1.6 (19.73) | -6.0 (22.01) | -6.1 (16.80)
  Week 19 (n= 164, 96, 98): number analyzed (Participants) | 164 | 96 | 98
  Week 19 (n= 164, 96, 98) | -0.8 (18.30) | -0.8 (21.70) | -5.4 (19.52)
  Week 23 (n= 134, 86, 75): number analyzed (Participants) | 134 | 86 | 75
  Week 23 (n= 134, 86, 75) | -2.8 (19.44) | -2.6 (22.00) | -3.7 (16.28)
  Week 25 (n= 144, 97, 75): number analyzed (Participants) | 144 | 97 | 75
  Week 25 (n= 144, 97, 75) | 1.3 (17.39) | -3.3 (17.70) | -4.2 (16.52)
  Week 31 (n= 123, 92, 51): number analyzed (Participants) | 123 | 92 | 51
  Week 31 (n= 123, 92, 51) | 2.5 (17.40) | 1.5 (21.47) | 2.0 (15.51)
  Week 37 (n= 116, 88, 48): number analyzed (Participants) | 116 | 88 | 48
  Week 37 (n= 116, 88, 48) | 3.2 (18.44) | -0.2 (21.18) | -1.9 (15.11)
  Week 43 (n= 103, 74, 44): number analyzed (Participants) | 103 | 74 | 44
  Week 43 (n= 103, 74, 44) | 3.5 (18.28) | -0.5 (23.04) | -0.9 (15.59)
  Week 49 (n= 97, 70, 40): number analyzed (Participants) | 97 | 70 | 40
  Week 49 (n= 97, 70, 40) | 2.7 (16.52) | 0.6 (21.95) | -0.4 (15.78)
  Week 55 (n= 86, 66, 34): number analyzed (Participants) | 86 | 66 | 34
  Week 55 (n= 86, 66, 34) | 1.8 (14.26) | -2.4 (22.01) | 0.7 (13.03)
  Week 61 (n= 85, 61, 31): number analyzed (Participants) | 85 | 61 | 31
  Week 61 (n= 85, 61, 31) | 1.6 (16.29) | -3.6 (20.78) | 0.8 (11.25)
  Week 67 (n= 76, 61, 29): number analyzed (Participants) | 76 | 61 | 29
  Week 67 (n= 76, 61, 29) | 2.1 (17.49) | -2.9 (21.35) | -6.6 (15.17)
  Week 73 (n= 67, 54, 19): number analyzed (Participants) | 67 | 54 | 19
  Week 73 (n= 67, 54, 19) | 0.1 (19.11) | -4.5 (21.76) | -3.5 (16.97)
  Week 79 (n= 67, 54, 21): number analyzed (Participants) | 67 | 54 | 21
  Week 79 (n= 67, 54, 21) | -0.1 (14.40) | -4.8 (20.51) | -0.8 (14.65)
  Week 85 (n= 68, 51, 18): number analyzed (Participants) | 68 | 51 | 18
  Week 85 (n= 68, 51, 18) | 2.8 (16.64) | -3.3 (22.37) | 0.0 (10.69)
  Week 91 (n= 62, 53, 16): number analyzed (Participants) | 62 | 53 | 16
  Week 91 (n= 62, 53, 16) | 0.9 (17.08) | -3.9 (20.78) | 0.5 (12.72)
  Week 97 (n= 58, 49, 17): number analyzed (Participants) | 58 | 49 | 17
  Week 97 (n= 58, 49, 17) | 0.9 (17.01) | -5.1 (23.06) | -2.9 (12.13)
  Week 103 (n= 53, 46, 17): number analyzed (Participants) | 53 | 46 | 17
  Week 103 (n= 53, 46, 17) | 2.2 (17.61) | -9.8 (19.03) | 0.0 (13.50)
  Week 109 (n= 44, 39, 14): number analyzed (Participants) | 44 | 39 | 14
  Week 109 (n= 44, 39, 14) | 2.8 (16.56) | -3.8 (23.17) | -2.4 (14.03)
  Week 115 (n= 44, 36, 17): number analyzed (Participants) | 44 | 36 | 17
  Week 115 (n= 44, 36, 17) | 0.6 (15.50) | -6.9 (22.76) | -0.5 (11.59)
  Week 121 (n= 44, 39, 16): number analyzed (Participants) | 44 | 39 | 16
  Week 121 (n= 44, 39, 16) | 1.1 (19.90) | -1.5 (19.20) | -3.1 (15.18)
  Week 127 (n= 47, 36, 17): number analyzed (Participants) | 47 | 36 | 17
  Week 127 (n= 47, 36, 17) | 0.9 (20.06) | -1.9 (22.37) | 1.5 (12.92)
  Week 133 (n= 29, 31, 11): number analyzed (Participants) | 29 | 31 | 11
  Week 133 (n= 29, 31, 11) | 3.2 (20.70) | -2.4 (25.11) | 3.8 (13.10)
  Week 139 (n= 20, 19, 6): number analyzed (Participants) | 20 | 19 | 6
  Week 139 (n= 20, 19, 6) | 0.0 (18.73) | -4.4 (17.43) | 5.6 (15.52)
  Week 145 (n= 14, 14, 6): number analyzed (Participants) | 14 | 14 | 6
  Week 145 (n= 14, 14, 6) | 0.6 (25.42) | -8.9 (8.93) | -4.2 (17.28)
  Week 151 (n= 7, 7, 1): number analyzed (Participants) | 7 | 7 | 1
  Week 151 (n= 7, 7, 1) | 3.6 (9.45) | -13.1 (9.45) | 8.3 (NA) — No SD calculated; only one patient analyzed
  Week 157 (n= 1, 3, 0): number analyzed (Participants) | 1 | 3 | 0
  Week 157 (n= 1, 3, 0) | 0.0 (NA) — No SD calculated; only one patient analyzed | -16.7 (8.33) |

11. Secondary Outcome: Mean Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Social Functioning
Description: as for outcome 10
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Points on EORTC scale
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 316 | 314 | 315
Points on EORTC scale
  Week 5 (n= 233, 183, 221): number analyzed (Participants) | 233 | 183 | 221
  Week 5 (n= 233, 183, 221) | -1.2 (21.99) | -4.6 (21.76) | -1.6 (21.59)
  Week 7 (n= 239, 183, 218): number analyzed (Participants) | 239 | 183 | 218
  Week 7 (n= 239, 183, 218) | -0.1 (20.58) | -5.8 (21.81) | -0.2 (21.79)
  Week 11 (n= 201, 112, 163): number analyzed (Participants) | 201 | 112 | 163
  Week 11 (n= 201, 112, 163) | -0.6 (22.32) | -5.1 (22.02) | -3.4 (21.53)
  Week 13 (n= 195, 106, 130): number analyzed (Participants) | 195 | 106 | 130
  Week 13 (n= 195, 106, 130) | 0.6 (22.73) | -3.6 (20.57) | -2.2 (24.41)
  Week 17 (n= 158, 84, 104): number analyzed (Participants) | 158 | 84 | 104
  Week 17 (n= 158, 84, 104) | -0.9 (22.28) | -4.4 (25.10) | -2.9 (18.06)
  Week 19 (n= 164, 96, 98): number analyzed (Participants) | 164 | 96 | 98
  Week 19 (n= 164, 96, 98) | 1.4 (21.40) | -1.7 (23.13) | -1.3 (24.71)
  Week 23 (n= 134, 86, 75): number analyzed (Participants) | 134 | 86 | 75
  Week 23 (n= 134, 86, 75) | -0.1 (19.87) | -1.2 (23.40) | -4.2 (21.94)
  Week 25 (n= 144, 97, 75): number analyzed (Participants) | 144 | 97 | 75
  Week 25 (n= 144, 97, 75) | 1.2 (19.77) | -3.4 (21.37) | -1.3 (25.23)
  Week 31 (n= 123, 92, 51): number analyzed (Participants) | 123 | 92 | 51
  Week 31 (n= 123, 92, 51) | 3.5 (16.84) | 0.2 (20.30) | 3.6 (22.68)
  Week 37 (n= 116, 88, 48): number analyzed (Participants) | 116 | 88 | 48
  Week 37 (n= 116, 88, 48) | 1.6 (18.12) | 1.1 (22.71) | 3.1 (18.40)
  Week 43 (n= 103, 74, 44): number analyzed (Participants) | 103 | 74 | 44
  Week 43 (n= 103, 74, 44) | -0.2 (20.68) | 2.9 (21.43) | 4.2 (22.77)
  Week 49 (n= 97, 70, 40): number analyzed (Participants) | 97 | 70 | 40
  Week 49 (n= 97, 70, 40) | 2.4 (17.35) | 3.1 (19.92) | 6.3 (18.37)
  Week 55 (n= 86, 66, 34): number analyzed (Participants) | 86 | 66 | 34
  Week 55 (n= 86, 66, 34) | 0.6 (19.21) | 0.0 (21.68) | 5.9 (17.83)
  Week 61 (n= 85, 61, 31): number analyzed (Participants) | 85 | 61 | 31
  Week 61 (n= 85, 61, 31) | 2.7 (16.44) | -0.5 (22.76) | 5.9 (17.51)
  Week 67 (n= 76, 61, 29): number analyzed (Participants) | 76 | 61 | 29
  Week 67 (n= 76, 61, 29) | 1.8 (16.46) | -0.8 (24.80) | -2.3 (17.66)
  Week 73 (n= 67, 54, 19): number analyzed (Participants) | 67 | 54 | 19
  Week 73 (n= 67, 54, 19) | 1.5 (17.58) | -2.5 (17.85) | -8.8 (18.73)
  Week 79 (n= 67, 54, 21): number analyzed (Participants) | 67 | 54 | 21
  Week 79 (n= 67, 54, 21) | 1.2 (14.01) | -3.4 (24.31) | 0.8 (3.64)
  Week 85 (n= 68, 51, 18): number analyzed (Participants) | 68 | 51 | 18
  Week 85 (n= 68, 51, 18) | 1.0 (13.77) | -7.5 (21.68) | -1.9 (7.86)
  Week 91 (n= 62, 53, 16): number analyzed (Participants) | 62 | 53 | 16
  Week 91 (n= 62, 53, 16) | -0.8 (17.96) | -5.7 (24.23) | 1.0 (4.17)
  Week 97 (n= 58, 49, 17): number analyzed (Participants) | 58 | 49 | 17
  Week 97 (n= 58, 49, 17) | -0.3 (16.95) | -2.7 (22.14) | 0.0 (0.00)
  Week 103 (n= 53, 46, 17): number analyzed (Participants) | 53 | 46 | 17
  Week 103 (n= 53, 46, 17) | -0.6 (17.28) | -4.3 (22.62) | -1.0 (4.04)
  Week 109 (n= 44, 39, 14): number analyzed (Participants) | 44 | 39 | 14
  Week 109 (n= 44, 39, 14) | 4.2 (15.72) | -2.6 (20.43) | -3.6 (9.65)
  Week 115 (n= 44, 36, 17): number analyzed (Participants) | 44 | 36 | 17
  Week 115 (n= 44, 36, 17) | 3.8 (18.63) | -2.3 (25.56) | 0.0 (5.89)
  Week 121 (n= 44, 39, 16): number analyzed (Participants) | 44 | 39 | 16
  Week 121 (n= 44, 39, 16) | 3.4 (19.88) | -3.0 (25.33) | -1.0 (4.17)
  Week 127 (n= 47, 36, 17): number analyzed (Participants) | 47 | 36 | 17
  Week 127 (n= 47, 36, 17) | 3.5 (18.37) | -2.3 (22.24) | 2.0 (5.54)
  Week 133 (n= 29, 31, 11): number analyzed (Participants) | 29 | 31 | 11
  Week 133 (n= 29, 31, 11) | 0.6 (15.74) | -2.2 (26.44) | 3.0 (10.05)
  Week 139 (n= 20, 19, 6): number analyzed (Participants) | 20 | 19 | 6
  Week 139 (n= 20, 19, 6) | 4.2 (10.64) | -4.4 (19.12) | 2.8 (16.39)
  Week 145 (n= 14, 14, 6): number analyzed (Participants) | 14 | 14 | 6
  Week 145 (n= 14, 14, 6) | -8.3 (26.75) | -11.9 (16.57) | 2.8 (16.39)
  Week 151 (n= 7, 7, 1): number analyzed (Participants) | 7 | 7 | 1
  Week 151 (n= 7, 7, 1) | 7.1 (23.29) | -9.5 (16.27) | 0 (NA) — No SD calculated; only one patient analyzed
  Week 157 (n= 1, 3, 0): number analyzed (Participants) | 1 | 3 | 0
  Week 157 (n= 1, 3, 0) | 0.0 (NA) — No SD calculated; only one patient analyzed | -22.2 (19.25) |

12. Secondary Outcome: Mean Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Cognitive Functioning
Description: as for outcome 10
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Points on EORTC scale
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 316 | 314 | 315
Points on EORTC scale
  Week 5 (n= 233, 183, 221): number analyzed (Participants) | 233 | 183 | 221
  Week 5 (n= 233, 183, 221) | 0.1 (12.28) | -2.1 (16.49) | -0.2 (13.99)
  Week 7 (n= 239, 183, 218): number analyzed (Participants) | 239 | 183 | 218
  Week 7 (n= 239, 183, 218) | -1.7 (12.80) | -3.6 (16.26) | -1.5 (13.36)
  Week 11 (n= 201, 112, 163): number analyzed (Participants) | 201 | 112 | 163
  Week 11 (n= 201, 112, 163) | -1.7 (13.27) | -0.1 (16.67) | -4.7 (15.33)
  Week 13 (n= 195, 106, 130): number analyzed (Participants) | 195 | 106 | 130
  Week 13 (n= 195, 106, 130) | -0.9 (13.45) | -0.3 (14.36) | -2.3 (14.64)
  Week 17 (n= 158, 84, 104): number analyzed (Participants) | 158 | 84 | 104
  Week 17 (n= 158, 84, 104) | -0.9 (12.79) | -3.6 (19.37) | -2.4 (13.43)
  Week 19 (n= 164, 96, 98): number analyzed (Participants) | 164 | 96 | 98
  Week 19 (n= 164, 96, 98) | -1.9 (13.99) | -1.0 (17.07) | -2.2 (13.39)
  Week 23 (n= 134, 86, 75): number analyzed (Participants) | 134 | 86 | 75
  Week 23 (n= 134, 86, 75) | -0.6 (13.31) | -4.5 (21.61) | -5.6 (14.58)
  Week 25 (n= 144, 97, 75): number analyzed (Participants) | 144 | 97 | 75
  Week 25 (n= 144, 97, 75) | -1.2 (12.72) | -4.8 (20.26) | -2.4 (12.46)
  Week 31 (n= 123, 92, 51): number analyzed (Participants) | 123 | 92 | 51
  Week 31 (n= 123, 92, 51) | 1.1 (12.40) | -1.6 (17.13) | -3.3 (12.48)
  Week 37 (n= 116, 88, 48): number analyzed (Participants) | 116 | 88 | 48
  Week 37 (n= 116, 88, 48) | 1.6 (11.42) | -2.8 (17.91) | -5.6 (15.88)
  Week 43 (n= 103, 74, 44): number analyzed (Participants) | 103 | 74 | 44
  Week 43 (n= 103, 74, 44) | -1.6 (15.40) | -2.9 (13.89) | 0.0 (11.37)
  Week 49 (n= 97, 70, 40): number analyzed (Participants) | 97 | 70 | 40
  Week 49 (n= 97, 70, 40) | -1.2 (12.32) | -1.2 (15.10) | 0.4 (12.22)
  Week 55 (n= 86, 66, 34): number analyzed (Participants) | 86 | 66 | 34
  Week 55 (n= 86, 66, 34) | 0.4 (13.52) | -2.8 (14.79) | -2.5 (12.40)
  Week 61 (n= 85, 61, 31): number analyzed (Participants) | 85 | 61 | 31
  Week 61 (n= 85, 61, 31) | 0.0 (14.09) | -1.6 (15.12) | -3.2 (15.76)
  Week 67 (n= 76, 61, 29): number analyzed (Participants) | 76 | 61 | 29
  Week 67 (n= 76, 61, 29) | -1.3 (13.27) | -3.0 (17.35) | -7.5 (16.42)
  Week 73 (n= 67, 54, 19): number analyzed (Participants) | 67 | 54 | 19
  Week 73 (n= 67, 54, 19) | -2.2 (11.20) | -4.9 (19.86) | -6.1 (11.40)
  Week 79 (n= 67, 54, 21): number analyzed (Participants) | 67 | 54 | 21
  Week 79 (n= 67, 54, 21) | -0.2 (12.48) | -4.6 (20.58) | -4.8 (13.06)
  Week 85 (n= 68, 51, 18): number analyzed (Participants) | 68 | 51 | 18
  Week 85 (n= 68, 51, 18) | -1.5 (12.79) | -4.2 (17.90) | -2.8 (13.10)
  Week 91 (n= 62, 53, 16): number analyzed (Participants) | 62 | 53 | 16
  Week 91 (n= 62, 53, 16) | -0.5 (12.06) | -4.7 (19.44) | -1.0 (9.56)
  Week 97 (n= 58, 49, 17): number analyzed (Participants) | 58 | 49 | 17
  Week 97 (n= 58, 49, 17) | -3.2 (14.12) | -3.7 (13.72) | -2.0 (10.00)
  Week 103 (n= 53, 46, 17): number analyzed (Participants) | 53 | 46 | 17
  Week 103 (n= 53, 46, 17) | -2.5 (15.81) | -5.8 (23.63) | -5.9 (15.52)
  Week 109 (n= 44, 39, 14): number analyzed (Participants) | 44 | 39 | 14
  Week 109 (n= 44, 39, 14) | 1.1 (10.42) | -3.8 (19.29) | -1.2 (7.91)
  Week 115 (n= 44, 36, 17): number analyzed (Participants) | 44 | 36 | 17
  Week 115 (n= 44, 36, 17) | 0.4 (9.84) | -3.7 (15.49) | -2.0 (10.00)
  Week 121 (n= 44, 39, 16): number analyzed (Participants) | 44 | 39 | 16
  Week 121 (n= 44, 39, 16) | -1.1 (14.56) | -7.7 (15.22) | -1.0 (9.56)
  Week 127 (n= 47, 36, 17): number analyzed (Participants) | 47 | 36 | 17
  Week 127 (n= 47, 36, 17) | -2.8 (17.83) | -3.2 (13.10) | -1.0 (13.78)
  Week 133 (n= 29, 31, 11): number analyzed (Participants) | 29 | 31 | 11
  Week 133 (n= 29, 31, 11) | -4.6 (22.67) | -3.8 (13.41) | 1.5 (8.99)
  Week 139 (n= 20, 19, 6): number analyzed (Participants) | 20 | 19 | 6
  Week 139 (n= 20, 19, 6) | -3.3 (6.84) | -6.1 (11.40) | 5.6 (8.61)
  Week 145 (n= 14, 14, 6): number analyzed (Participants) | 14 | 14 | 6
  Week 145 (n= 14, 14, 6) | -11.9 (29.55) | -4.8 (12.10) | -5.6 (17.21)
  Week 151 (n= 7, 7, 1): number analyzed (Participants) | 7 | 7 | 1
  Week 151 (n= 7, 7, 1) | -2.4 (11.50) | -7.1 (13.11) | 16.7 (NA) — No SD calculated; only one patient analyzed
  Week 157 (n= 1, 3, 0): number analyzed (Participants) | 1 | 3 | 0
  Week 157 (n= 1, 3, 0) | 0.0 (NA) — No SD calculated; only one patient analyzed | -11.1 (9.62) |

13. Secondary Outcome: Mean Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Emotional Functioning
Description: as for outcome 10
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Points on EORTC scale
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 316 | 314 | 315
Points on EORTC scale
  Week 5 (n= 233, 183, 221): number analyzed (Participants) | 233 | 183 | 221
  Week 5 (n= 233, 183, 221) | 4.6 (15.91) | 2.5 (16.44) | 3.7 (17.21)
  Week 7 (n= 239, 183, 218): number analyzed (Participants) | 239 | 183 | 218
  Week 7 (n= 239, 183, 218) | 4.0 (16.82) | 2.0 (18.10) | 3.1 (17.39)
  Week 11 (n= 201, 112, 163): number analyzed (Participants) | 201 | 112 | 163
  Week 11 (n= 201, 112, 163) | 5.3 (14.84) | 3.7 (15.57) | 2.0 (18.89)
  Week 13 (n= 195, 106, 130): number analyzed (Participants) | 195 | 106 | 130
  Week 13 (n= 195, 106, 130) | 3.8 (15.99) | 4.3 (17.53) | 2.9 (18.03)
  Week 17 (n= 158, 84, 104): number analyzed (Participants) | 158 | 84 | 104
  Week 17 (n= 158, 84, 104) | 5.6 (16.54) | 4.2 (18.81) | 4.9 (15.86)
  Week 19 (n= 164, 96, 98): number analyzed (Participants) | 164 | 96 | 98
  Week 19 (n= 164, 96, 98) | 5.8 (16.26) | 6.2 (19.01) | 6.5 (18.27)
  Week 23 (n= 134, 86, 75): number analyzed (Participants) | 134 | 86 | 75
  Week 23 (n= 134, 86, 75) | 6.1 (17.04) | 4.5 (20.20) | 3.7 (18.85)
  Week 25 (n= 144, 97, 75): number analyzed (Participants) | 144 | 97 | 75
  Week 25 (n= 144, 97, 75) | 6.6 (16.31) | 2.1 (19.69) | 5.9 (17.15)
  Week 31 (n= 123, 92, 51): number analyzed (Participants) | 123 | 92 | 51
  Week 31 (n= 123, 92, 51) | 8.3 (15.57) | 4.7 (15.64) | 9.2 (16.69)
  Week 37 (n= 116, 88, 48): number analyzed (Participants) | 116 | 88 | 48
  Week 37 (n= 116, 88, 48) | 9.6 (15.60) | 6.8 (17.98) | 5.9 (16.75)
  Week 43 (n= 103, 74, 44): number analyzed (Participants) | 103 | 74 | 44
  Week 43 (n= 103, 74, 44) | 6.7 (18.89) | 7.5 (18.36) | 6.1 (14.86)
  Week 49 (n= 97, 70, 40): number analyzed (Participants) | 97 | 70 | 40
  Week 49 (n= 97, 70, 40) | 5.8 (18.61) | 7.1 (19.67) | 8.1 (15.50)
  Week 55 (n= 86, 66, 34): number analyzed (Participants) | 86 | 66 | 34
  Week 55 (n= 86, 66, 34) | 8.1 (18.57) | 8.3 (16.79) | 12.3 (15.11)
  Week 61 (n= 85, 61, 31): number analyzed (Participants) | 85 | 61 | 31
  Week 61 (n= 85, 61, 31) | 7.9 (18.54) | 7.9 (22.69) | 9.9 (14.82)
  Week 67 (n= 76, 61, 29): number analyzed (Participants) | 76 | 61 | 29
  Week 67 (n= 76, 61, 29) | 7.8 (19.97) | 7.1 (20.52) | 3.7 (15.36)
  Week 73 (n= 67, 54, 19): number analyzed (Participants) | 67 | 54 | 19
  Week 73 (n= 67, 54, 19) | 8.0 (18.66) | 4.5 (18.29) | 4.8 (10.51)
  Week 79 (n= 67, 54, 21): number analyzed (Participants) | 67 | 54 | 21
  Week 79 (n= 67, 54, 21) | 7.6 (19.56) | 2.9 (23.36) | 6.7 (10.41)
  Week 85 (n= 68, 51, 18): number analyzed (Participants) | 68 | 51 | 18
  Week 85 (n= 68, 51, 18) | 6.4 (16.55) | 3.3 (21.09) | 7.9 (12.61)
  Week 91 (n= 62, 53, 16): number analyzed (Participants) | 62 | 53 | 16
  Week 91 (n= 62, 53, 16) | 9.1 (17.77) | 4.7 (20.25) | 3.6 (12.53)
  Week 97 (n= 58, 49, 17): number analyzed (Participants) | 58 | 49 | 17
  Week 97 (n= 58, 49, 17) | 5.3 (17.78) | 3.9 (21.05) | 3.9 (14.47)
  Week 103 (n= 53, 46, 17): number analyzed (Participants) | 53 | 46 | 17
  Week 103 (n= 53, 46, 17) | 6.6 (19.50) | 1.4 (23.46) | 4.4 (12.88)
  Week 109 (n= 44, 39, 14): number analyzed (Participants) | 44 | 39 | 14
  Week 109 (n= 44, 39, 14) | 8.3 (17.33) | 4.1 (22.61) | 12.5 (11.20)
  Week 115 (n= 44, 36, 17): number analyzed (Participants) | 44 | 36 | 17
  Week 115 (n= 44, 36, 17) | 8.1 (21.15) | 6.0 (21.23) | 10.3 (10.84)
  Week 121 (n= 44, 39, 16): number analyzed (Participants) | 44 | 39 | 16
  Week 121 (n= 44, 39, 16) | 8.3 (20.01) | 4.5 (21.36) | 9.4 (7.98)
  Week 127 (n= 47, 36, 17): number analyzed (Participants) | 47 | 36 | 17
  Week 127 (n= 47, 36, 17) | 10.6 (17.61) | 7.2 (21.19) | 8.3 (13.50)
  Week 133 (n= 29, 31, 11): number analyzed (Participants) | 29 | 31 | 11
  Week 133 (n= 29, 31, 11) | 7.5 (19.46) | 8.3 (19.48) | 9.1 (7.87)
  Week 139 (n= 20, 19, 6): number analyzed (Participants) | 20 | 19 | 6
  Week 139 (n= 20, 19, 6) | 9.6 (11.87) | 9.2 (16.87) | 11.1 (10.09)
  Week 145 (n= 14, 14, 6): number analyzed (Participants) | 14 | 14 | 6
  Week 145 (n= 14, 14, 6) | 2.4 (18.32) | 6.0 (15.82) | 11.1 (10.09)
  Week 151 (n= 7, 7, 1): number analyzed (Participants) | 7 | 7 | 1
  Week 151 (n= 7, 7, 1) | 17.9 (16.27) | -2.4 (22.93) | 16.7 (NA) — No SD calculated; only one patient analyzed
  Week 157 (n= 1, 3, 0): number analyzed (Participants) | 1 | 3 | 0
  Week 157 (n= 1, 3, 0) | 16.7 (NA) — No SD calculated; only one patient analyzed | -11.1 (17.35) |

14. Secondary Outcome: Mean Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Role Functioning
Description: as for outcome 10
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Points on EORTC scale
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 316 | 314 | 315
Points on EORTC scale
  Week 5 (n= 233, 183, 221): number analyzed (Participants) | 233 | 183 | 221
  Week 5 (n= 233, 183, 221) | -4.1 (23.71) | -6.8 (24.90) | -4.4 (21.18)
  Week 7 (n= 239, 183, 218): number analyzed (Participants) | 239 | 183 | 218
  Week 7 (n= 239, 183, 218) | -3.6 (24.21) | -11.6 (28.25) | -4.9 (22.44)
  Week 11 (n= 201, 112, 163): number analyzed (Participants) | 201 | 112 | 163
  Week 11 (n= 201, 112, 163) | -3.2 (24.46) | -9.7 (28.97) | -6.1 (24.56)
  Week 13 (n= 195, 106, 130): number analyzed (Participants) | 195 | 106 | 130
  Week 13 (n= 195, 106, 130) | -3.1 (24.15) | -8.3 (25.33) | -6.9 (25.65)
  Week 17 (n= 158, 84, 104): number analyzed (Participants) | 158 | 84 | 104
  Week 17 (n= 158, 84, 104) | -3.2 (26.14) | -11.1 (27.05) | -6.3 (20.27)
  Week 19 (n= 164, 96, 98): number analyzed (Participants) | 164 | 96 | 98
  Week 19 (n= 164, 96, 98) | -1.3 (24.56) | -4.3 (25.04) | -6.1 (24.80)
  Week 23 (n= 134, 86, 75): number analyzed (Participants) | 134 | 86 | 75
  Week 23 (n= 134, 86, 75) | -2.6 (25.76) | -6.4 (24.14) | -8.4 (24.56)
  Week 25 (n= 144, 97, 75): number analyzed (Participants) | 144 | 97 | 75
  Week 25 (n= 144, 97, 75) | 0.7 (21.13) | -7.7 (23.70) | -7.8 (23.78)
  Week 31 (n= 123, 92, 51): number analyzed (Participants) | 123 | 92 | 51
  Week 31 (n= 123, 92, 51) | -0.7 (21.38) | -3.1 (24.82) | -3.9 (23.24)
  Week 37 (n= 116, 88, 48): number analyzed (Participants) | 116 | 88 | 48
  Week 37 (n= 116, 88, 48) | 1.6 (22.94) | -3.2 (26.37) | -3.1 (21.92)
  Week 43 (n= 103, 74, 44): number analyzed (Participants) | 103 | 74 | 44
  Week 43 (n= 103, 74, 44) | 1.0 (20.85) | -3.4 (26.46) | -1.1 (19.49)
  Week 49 (n= 97, 70, 40): number analyzed (Participants) | 97 | 70 | 40
  Week 49 (n= 97, 70, 40) | 1.7 (20.62) | -1.2 (21.67) | -2.1 (21.08)
  Week 55 (n= 86, 66, 34): number analyzed (Participants) | 86 | 66 | 34
  Week 55 (n= 86, 66, 34) | 1.6 (20.07) | -4.8 (21.03) | 1.0 (16.89)
  Week 61 (n= 85, 61, 31): number analyzed (Participants) | 85 | 61 | 31
  Week 61 (n= 85, 61, 31) | 0.4 (19.58) | -3.0 (24.82) | 1.1 (21.05)
  Week 67 (n= 76, 61, 29): number analyzed (Participants) | 76 | 61 | 29
  Week 67 (n= 76, 61, 29) | 0.7 (19.33) | -4.6 (25.84) | -1.7 (17.45)
  Week 73 (n= 67, 54, 19): number analyzed (Participants) | 67 | 54 | 19
  Week 73 (n= 67, 54, 19) | 0.5 (19.24) | -5.6 (26.70) | -0.9 (17.10)
  Week 79 (n= 67, 54, 21): number analyzed (Participants) | 67 | 54 | 21
  Week 79 (n= 67, 54, 21) | -0.7 (18.45) | -8.3 (27.99) | -2.4 (12.12)
  Week 85 (n= 68, 51, 18): number analyzed (Participants) | 68 | 51 | 18
  Week 85 (n= 68, 51, 18) | -2.2 (16.26) | -9.8 (28.90) | 0.9 (12.09)
  Week 91 (n= 62, 53, 16): number analyzed (Participants) | 62 | 53 | 16
  Week 91 (n= 62, 53, 16) | 1.1 (22.76) | -10.7 (29.25) | 2.1 (13.44)
  Week 97 (n= 58, 49, 17): number analyzed (Participants) | 58 | 49 | 17
  Week 97 (n= 58, 49, 17) | 0.6 (23.77) | -7.5 (26.80) | 0.0 (13.18)
  Week 103 (n= 53, 46, 17): number analyzed (Participants) | 53 | 46 | 17
  Week 103 (n= 53, 46, 17) | -0.6 (26.95) | -9.8 (23.46) | 2.0 (10.00)
  Week 109 (n= 44, 39, 14): number analyzed (Participants) | 44 | 39 | 14
  Week 109 (n= 44, 39, 14) | 1.1 (21.98) | -5.6 (22.73) | 4.8 (10.19)
  Week 115 (n= 44, 36, 17): number analyzed (Participants) | 44 | 36 | 17
  Week 115 (n= 44, 36, 17) | 1.1 (22.27) | -10.6 (28.77) | 2.0 (11.61)
  Week 121 (n= 44, 39, 16): number analyzed (Participants) | 44 | 39 | 16
  Week 121 (n= 44, 39, 16) | 0.4 (28.41) | -8.1 (26.73) | 2.1 (14.75)
  Week 127 (n= 47, 36, 17): number analyzed (Participants) | 47 | 36 | 17
  Week 127 (n= 47, 36, 17) | 1.4 (24.03) | -6.0 (26.17) | 1.0 (7.15)
  Week 133 (n= 29, 31, 11): number analyzed (Participants) | 29 | 31 | 11
  Week 133 (n= 29, 31, 11) | 1.1 (34.48) | -4.3 (24.33) | -1.5 (11.68)
  Week 139 (n= 20, 19, 6): number analyzed (Participants) | 20 | 19 | 6
  Week 139 (n= 20, 19, 6) | -5.8 (9.79) | -8.8 (18.73) | 8.3 (13.94)
  Week 145 (n= 14, 14, 6): number analyzed (Participants) | 14 | 14 | 6
  Week 145 (n= 14, 14, 6) | -6.0 (34.96) | -10.7 (16.80) | 0.0 (23.57)
  Week 151 (n= 7, 7, 1): number analyzed (Participants) | 7 | 7 | 1
  Week 151 (n= 7, 7, 1) | 7.1 (26.97) | -14.3 (17.82) | 0.0 (NA) — No SD calculated; only one patient analyzed
  Week 157 (n= 1, 3, 0): number analyzed (Participants) | 1 | 3 | 0
  Week 157 (n= 1, 3, 0) | 0.0 (NA) — No SD calculated; only one patient analyzed | -11.1 (19.25) |

15. Secondary Outcome: Mean Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Physical Functioning
Description: as for outcome 10
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Points on EORTC scale
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab
Number analyzed (Participants) | 316 | 314 | 315
Points on EORTC scale
  Week 5 (n= 233, 183, 221): number analyzed (Participants) | 233 | 183 | 221
  Week 5 (n= 233, 183, 221) | -2.6 (13.62) | -4.9 (14.52) | -5.2 (14.09)
  Week 7 (n= 239, 183, 218): number analyzed (Participants) | 239 | 183 | 218
  Week 7 (n= 239, 183, 218) | -2.4 (14.53) | -5.3 (14.92) | -5.1 (14.69)
  Week 11 (n= 201, 112, 163): number analyzed (Participants) | 201 | 112 | 163
  Week 11 (n= 201, 112, 163) | -2.4 (16.14) | -5.6 (13.76) | -6.3 (14.72)
  Week 13 (n= 195, 106, 130): number analyzed (Participants) | 195 | 106 | 130
  Week 13 (n= 195, 106, 130) | -1.7 (15.79) | -4.3 (14.11) | -5.0 (17.47)
  Week 17 (n= 158, 84, 104): number analyzed (Participants) | 158 | 84 | 104
  Week 17 (n= 158, 84, 104) | -1.4 (15.82) | -6.7 (17.27) | -3.7 (13.46)
  Week 19 (n= 164, 96, 98): number analyzed (Participants) | 164 | 96 | 98
  Week 19 (n= 164, 96, 98) | 0.4 (14.14) | -3.7 (14.34) | -4.3 (17.70)
  Week 23 (n= 134, 86, 75): number analyzed (Participants) | 134 | 86 | 75
  Week 23 (n= 134, 86, 75) | 0.9 (13.87) | -4.0 (15.59) | -5.5 (15.04)
  Week 25 (n= 144, 97, 75): number analyzed (Participants) | 144 | 97 | 75
  Week 25 (n= 144, 97, 75) | 1.4 (11.02) | -4.2 (14.28) | -3.6 (16.19)
  Week 31 (n= 123, 92, 51): number analyzed (Participants) | 123 | 92 | 51
  Week 31 (n= 123, 92, 51) | 1.9 (11.60) | -2.4 (12.91) | -2.9 (14.62)
  Week 37 (n= 116, 88, 48): number analyzed (Participants) | 116 | 88 | 48
  Week 37 (n= 116, 88, 48) | 2.1 (13.57) | -0.8 (13.00) | -2.2 (13.71)
  Week 43 (n= 103, 74, 44): number analyzed (Participants) | 103 | 74 | 44
  Week 43 (n= 103, 74, 44) | 1.9 (13.16) | -0.5 (13.55) | -1.7 (12.71)
  Week 49 (n= 97, 70, 40): number analyzed (Participants) | 97 | 70 | 40
  Week 49 (n= 97, 70, 40) | 1.3 (12.08) | -0.1 (12.97) | 0.2 (12.31)
  Week 55 (n= 86, 66, 34): number analyzed (Participants) | 86 | 66 | 34
  Week 55 (n= 86, 66, 34) | 1.8 (11.68) | -2.9 (13.24) | 0.2 (10.57)
  Week 61 (n= 85, 61, 31): number analyzed (Participants) | 85 | 61 | 31
  Week 61 (n= 85, 61, 31) | 0.2 (11.65) | -2.1 (13.91) | -0.2 (11.35)
  Week 67 (n= 76, 61, 29): number analyzed (Participants) | 76 | 61 | 29
  Week 67 (n= 76, 61, 29) | 0.9 (12.44) | -1.7 (13.22) | -3.9 (10.62)
  Week 73 (n= 67, 54, 19): number analyzed (Participants) | 67 | 54 | 19
  Week 73 (n= 67, 54, 19) | 0.5 (14.38) | -3.5 (11.27) | -3.9 (7.80)
  Week 79 (n= 67, 54, 21): number analyzed (Participants) | 67 | 54 | 21
  Week 79 (n= 67, 54, 21) | -1.7 (7.99) | -4.3 (17.09) | -1.3 (6.54)
  Week 85 (n= 68, 51, 18): number analyzed (Participants) | 68 | 51 | 18
  Week 85 (n= 68, 51, 18) | -1.6 (12.86) | -3.5 (12.88) | -2.6 (6.11)
  Week 91 (n= 62, 53, 16): number analyzed (Participants) | 62 | 53 | 16
  Week 91 (n= 62, 53, 16) | -0.4 (13.27) | -4.2 (14.45) | 0.0 (0.00)
  Week 97 (n= 58, 49, 17): number analyzed (Participants) | 58 | 49 | 17
  Week 97 (n= 58, 49, 17) | -0.4 (13.79) | -4.4 (16.53) | -0.8 (4.00)
  Week 103 (n= 53, 46, 17): number analyzed (Participants) | 53 | 46 | 17
  Week 103 (n= 53, 46, 17) | -1.5 (17.18) | -5.4 (15.63) | -2.4 (7.05)
  Week 109 (n= 44, 39, 14): number analyzed (Participants) | 44 | 39 | 14
  Week 109 (n= 44, 39, 14) | 1.7 (14.74) | -1.2 (13.92) | -1.0 (3.56)
  Week 115 (n= 44, 36, 17): number analyzed (Participants) | 44 | 36 | 17
  Week 115 (n= 44, 36, 17) | 0.2 (14.20) | -2.0 (15.10) | -0.8 (3.23)
  Week 121 (n= 44, 39, 16): number analyzed (Participants) | 44 | 39 | 16
  Week 121 (n= 44, 39, 16) | -0.3 (15.77) | -3.4 (13.58) | -2.5 (5.37)
  Week 127 (n= 47, 36, 17): number analyzed (Participants) | 47 | 36 | 17
  Week 127 (n= 47, 36, 17) | 1.2 (17.21) | -3.0 (16.75) | -2.4 (5.75)
  Week 133 (n= 29, 31, 11): number analyzed (Participants) | 29 | 31 | 11
  Week 133 (n= 29, 31, 11) | 0.2 (23.33) | 0.4 (14.40) | -2.4 (6.16)
  Week 139 (n= 20, 19, 6): number analyzed (Participants) | 20 | 19 | 6
  Week 139 (n= 20, 19, 6) | 0.4 (7.94) | -3.9 (11.40) | -3.3 (5.58)
  Week 145 (n= 14, 14, 6): number analyzed (Participants) | 14 | 14 | 6
  Week 145 (n= 14, 14, 6) | -1.4 (27.94) | -6.7 (9.06) | -6.7 (8.43)
  Week 151 (n= 7, 7, 1): number analyzed (Participants) | 7 | 7 | 1
  Week 151 (n= 7, 7, 1) | 8.6 (17.52) | -9.5 (12.68) | 0.0 (NA) — No SD calculated; only one patient analyzed
  Week 157 (n= 1, 3, 0): number analyzed (Participants) | 1 | 3 | 0
  Week 157 (n= 1, 3, 0) | 0.0 (NA) — No SD calculated; only one patient analyzed | -17.8 (25.24) |

ADVERSE EVENTS:
Time Frame: All cause mortality was collected from date of randomization till death due to any cause (up to approximately 128 months) and Serious and Other Adverse events were collected from first dose till 30 days after last dose (up to approximately 128 months).
Description: All cause mortality data was collected for all the randomized participants and serious and other adverse events were collected for all the treated participants.
Arm/Group | Nivolumab | Nivolumab + Ipilimumab | Ipilimumab
All-Cause Mortality (participants affected / at risk) | 192/316 | 173/314 | 243/315
Serious Adverse Events (participants affected / at risk) | 187/313 | 249/313 | 205/311
Other Adverse Events (participants affected / at risk) | 302/313 | 302/313 | 302/311
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=313) | Nivolumab + Ipilimumab (N=313) | Ipilimumab (N=311)
Anaemia (Blood and lymphatic system disorders) | 5 | 4 | 5
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 0 | 1
Bicytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 4 | 1
Atrial flutter (Cardiac disorders) | 1 | 1 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 2
Cardiac failure (Cardiac disorders) | 0 | 2 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 2
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 1 | 0
Cor pulmonale (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Adrenal haemorrhage (Endocrine disorders) | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 3 | 7 | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 1 | 0
Endocrine disorder (Endocrine disorders) | 0 | 1 | 0
Glucocorticoid deficiency (Endocrine disorders) | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 6 | 0
Hypophysitis (Endocrine disorders) | 1 | 8 | 8
Hypopituitarism (Endocrine disorders) | 1 | 3 | 2
Hypothyroidism (Endocrine disorders) | 0 | 2 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 1
Lymphocytic hypophysitis (Endocrine disorders) | 0 | 1 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 1 | 0
Thyroiditis (Endocrine disorders) | 0 | 2 | 0
Diplopia (Eye disorders) | 1 | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 1
Uveitis (Eye disorders) | 1 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 5 | 7
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 2 | 2 | 1
Autoimmune colitis (Gastrointestinal disorders) | 1 | 0 | 1
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 6 | 33 | 29
Constipation (Gastrointestinal disorders) | 3 | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 8 | 40 | 26
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 2 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2
Intestinal perforation (Gastrointestinal disorders) | 0 | 2 | 1
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Intussusception (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 3
Lymphangiectasia intestinal (Gastrointestinal disorders) | 1 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 9 | 3
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 2 | 5
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 11 | 3
Accidental death (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 2
Catheter site discharge (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 2 | 0 | 0
Chills (General disorders) | 0 | 0 | 1
Death (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 6 | 2
General physical health deterioration (General disorders) | 3 | 10 | 4
Hyperthermia (General disorders) | 1 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 2 | 0
Malaise (General disorders) | 1 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0
Nodule (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 0 | 1
Pain (General disorders) | 3 | 4 | 2
Performance status decreased (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 4 | 30 | 12
Sudden cardiac death (General disorders) | 0 | 1 | 0
Sudden death (General disorders) | 2 | 2 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 3 | 6 | 2
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 2 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 2 | 5 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0
Hepatorenal failure (Hepatobiliary disorders) | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 5 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 7 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0 | 0
Abscess intestinal (Infections and infestations) | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Biliary sepsis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2 | 1
Bursitis infective (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 3 | 3 | 3
Citrobacter sepsis (Infections and infestations) | 1 | 0 | 0
Clostridium bacteraemia (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 2 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 1 | 1
Diverticulitis intestinal perforated (Infections and infestations) | 1 | 0 | 0
Encephalitis (Infections and infestations) | 1 | 1 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 2 | 1 | 2
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0
Febrile infection (Infections and infestations) | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 3 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 2 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1
Groin abscess (Infections and infestations) | 0 | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 2 | 2 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 1
Meningitis (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 2 | 0
Pneumonia (Infections and infestations) | 3 | 9 | 5
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 5 | 3 | 1
Septic shock (Infections and infestations) | 1 | 1 | 2
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 3 | 4
Urosepsis (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0
Osteoradionecrosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Cortisol decreased (Investigations) | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
General physical condition abnormal (Investigations) | 1 | 0 | 2
Hepatic enzyme increased (Investigations) | 1 | 3 | 0
Lipase increased (Investigations) | 0 | 2 | 0
Liver function test increased (Investigations) | 2 | 1 | 0
Transaminases increased (Investigations) | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 10 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 7 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Steroid diabetes (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Adenoid cystic carcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 3 | 3
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Desmoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Infected metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Intestinal metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 54 | 38 | 61
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 5
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 3
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 2 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Diabetic coma (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 1
Facial paralysis (Nervous system disorders) | 0 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Intracranial tumour haemorrhage (Nervous system disorders) | 1 | 0 | 1
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Medullary compression syndrome (Nervous system disorders) | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 1 | 0 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 2
Sensory disturbance (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Spinal claudication (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 3 | 4 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 3 | 0
Device breakage (Product Issues) | 1 | 0 | 1
Device loosening (Product Issues) | 0 | 1 | 0
Device malfunction (Product Issues) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 4 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 2
Delusion (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 10 | 4
Autoimmune nephritis (Renal and urinary disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 1 | 0
Immune-mediated nephritis (Renal and urinary disorders) | 1 | 0 | 0
Lower urinary tract symptoms (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 1 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 3 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Renal mass (Renal and urinary disorders) | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Ejaculation failure (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 3
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Hepatic hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 11 | 5
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Vasculitic ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Embolism (Vascular disorders) | 2 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 4 | 1
Inferior vena caval occlusion (Vascular disorders) | 0 | 1 | 0
Lymphorrhoea (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=313) | Nivolumab + Ipilimumab (N=313) | Ipilimumab (N=311)
Anaemia (Blood and lymphatic system disorders) | 35 | 41 | 43
Tachycardia (Cardiac disorders) | 6 | 16 | 13
Adrenal insufficiency (Endocrine disorders) | 4 | 16 | 7
Hyperthyroidism (Endocrine disorders) | 18 | 30 | 3
Hypophysitis (Endocrine disorders) | 5 | 20 | 9
Hypothyroidism (Endocrine disorders) | 38 | 68 | 17
Dry eye (Eye disorders) | 17 | 12 | 8
Vision blurred (Eye disorders) | 18 | 18 | 15
Abdominal distension (Gastrointestinal disorders) | 17 | 9 | 13
Abdominal pain (Gastrointestinal disorders) | 62 | 59 | 68
Abdominal pain upper (Gastrointestinal disorders) | 24 | 24 | 25
Colitis (Gastrointestinal disorders) | 9 | 21 | 15
Constipation (Gastrointestinal disorders) | 69 | 63 | 77
Diarrhoea (Gastrointestinal disorders) | 122 | 168 | 147
Dry mouth (Gastrointestinal disorders) | 28 | 34 | 17
Dyspepsia (Gastrointestinal disorders) | 17 | 12 | 14
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 19 | 13 | 14
Nausea (Gastrointestinal disorders) | 105 | 136 | 104
Vomiting (Gastrointestinal disorders) | 69 | 99 | 60
Asthenia (General disorders) | 47 | 50 | 29
Chest pain (General disorders) | 19 | 12 | 13
Chills (General disorders) | 23 | 35 | 20
Fatigue (General disorders) | 159 | 168 | 140
Influenza like illness (General disorders) | 31 | 28 | 25
Oedema peripheral (General disorders) | 39 | 39 | 45
Pain (General disorders) | 18 | 23 | 29
Pyrexia (General disorders) | 64 | 123 | 61
Conjunctivitis (Infections and infestations) | 5 | 19 | 6
Influenza (Infections and infestations) | 16 | 20 | 8
Nasopharyngitis (Infections and infestations) | 43 | 34 | 29
Rhinitis (Infections and infestations) | 20 | 26 | 10
Sinusitis (Infections and infestations) | 16 | 14 | 5
Upper respiratory tract infection (Infections and infestations) | 32 | 28 | 17
Urinary tract infection (Infections and infestations) | 16 | 23 | 9
Alanine aminotransferase increased (Investigations) | 25 | 69 | 18
Amylase increased (Investigations) | 23 | 33 | 17
Aspartate aminotransferase increased (Investigations) | 25 | 61 | 19
Blood alkaline phosphatase increased (Investigations) | 14 | 19 | 8
Blood creatinine increased (Investigations) | 7 | 25 | 15
Gamma-glutamyltransferase increased (Investigations) | 7 | 16 | 10
Lipase increased (Investigations) | 35 | 51 | 21
Weight decreased (Investigations) | 28 | 42 | 26
Decreased appetite (Metabolism and nutrition disorders) | 76 | 97 | 76
Dehydration (Metabolism and nutrition disorders) | 7 | 24 | 17
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 18 | 17
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 16 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 37 | 15
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 25 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 87 | 79 | 78
Back pain (Musculoskeletal and connective tissue disorders) | 58 | 46 | 53
Groin pain (Musculoskeletal and connective tissue disorders) | 17 | 5 | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 22 | 16 | 16
Muscular weakness (Musculoskeletal and connective tissue disorders) | 13 | 22 | 12
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 16 | 13 | 16
Myalgia (Musculoskeletal and connective tissue disorders) | 34 | 33 | 23
Neck pain (Musculoskeletal and connective tissue disorders) | 15 | 18 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 49 | 38 | 43
Dizziness (Nervous system disorders) | 33 | 43 | 30
Dysgeusia (Nervous system disorders) | 17 | 18 | 8
Headache (Nervous system disorders) | 79 | 82 | 78
Paraesthesia (Nervous system disorders) | 23 | 18 | 17
Anxiety (Psychiatric disorders) | 11 | 24 | 19
Depression (Psychiatric disorders) | 12 | 21 | 9
Insomnia (Psychiatric disorders) | 44 | 51 | 42
Cough (Respiratory, thoracic and mediastinal disorders) | 100 | 82 | 69
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 47 | 72 | 43
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 20 | 8 | 14
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 21 | 15 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 | 23 | 17
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 17 | 7
Actinic keratosis (Skin and subcutaneous tissue disorders) | 17 | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 28 | 30 | 19
Erythema (Skin and subcutaneous tissue disorders) | 25 | 16 | 14
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 12 | 22 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 92 | 126 | 135
Rash (Skin and subcutaneous tissue disorders) | 101 | 111 | 84
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 22 | 44 | 43
Skin lesion (Skin and subcutaneous tissue disorders) | 20 | 11 | 9
Vitiligo (Skin and subcutaneous tissue disorders) | 38 | 29 | 17
Hypertension (Vascular disorders) | 34 | 26 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.